CLINICAL TRIAL: NCT04292743
Title: A Phase I Dose Escalation Study of Eryaspase in Combination With Modified FOLFIRINOX in Locally Advanced and Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Eryaspase With Modified FOLFIRINOX in Advanced Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002008
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — eryaspase; folfirinox; Fluorouracil; Oxaliplatin; Irinotecan; Leucovorin

STUDY DESIGN:
Intervention Model Description: Dose escalation of Eryaspase in combination with FOLFIRINOX
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Eryaspase Dose level 0 (75 Units/kg) plus FOLFIRINOX (Experimental): Eryaspase 75 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion).
  mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
  Interventions: Biological: Eryaspase; Drug: FOLFIRINOX
- Eryaspase Dose level 1 (100 Units/kg) plus FOLFIRINOX (Experimental): Eryaspase 100 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion).
  mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
  Interventions: Biological: Eryaspase; Drug: FOLFIRINOX
- Eryaspase Dose Level -1 (50 Units/kg) plus FOLFIRINOX (Experimental): Eryaspase 50 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion).
  mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
  Interventions: Biological: Eryaspase; Drug: FOLFIRINOX
- Eryaspase Dose Level -2 (25 Units/kg) plus FOLFIRINOX (Experimental): Eryaspase 25 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion).
  mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
  Interventions: Biological: Eryaspase; Drug: FOLFIRINOX

INTERVENTIONS:
Biological: Eryaspase — intravenous administration of Eryaspase, starting dose 75 units/kg, dose escalation to 100 units/kg, dose reduction 50 units/kg and 25 units/kg
Drug: FOLFIRINOX — intravenous administration of FOLFIRINOX
  Other Names: 5-fluorouracil, oxaliplatin, Irinotecan, leucovorin

SUMMARY:
This will be a single-arm, multi-center, open-label phase 1 study. The standard 3+3 design will be used to determine the maximum tolerated dose (MTD) from 4 possible dose levels of Eryaspase in combination with mFOLFIRINOX. We hypothesize that the addition of Eryaspase to FOLFIRINOX (5-fluorouracil [5-FU], leucovorin, irinotecan, and oxaliplatin) will be safe and demonstrate preliminary signs of efficacy in patients with advanced pancreatic cancer. Safety assessments include adverse events, physical examination abnormalities, vital signs, and clinical laboratory tests (including blood chemistry, hematology, and coagulation panel).

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1 study of Eryaspase combination with FOLFIRINOX in patients with locally advanced or metastatic pancreatic adenocarcinoma. Subjects will undergo screening in order to determine eligibility.

The study will use a standard 3+3 method of dose escalation. Patients will be enrolled in cohorts of 3. Four dose levels are planned and include 25, 50, 75, and 100 mg of Eryaspase with reduced dose irinotecan. Subjects will be assigned to a dose level in the order of study entry with at least a 3-day stagger in enrollment between individual subjects. With the 3+3 design to be employed, doses are not escalated unless all patients receiving the current dose have been observed for at least 6 weeks and dose-limiting toxicities (DLTs) have been reported. The MTD is defined as the highest dose level where at most 1 of 6 patients experience a dose limiting toxicity (DLT). Three patients will be treated at dose level 0. If 0/3 experience a DLT, 3 new patients will be enrolled at the next higher dose level. If 1/3 experience a DLT, 3 additional patients will be enrolled at the same dose level. If 1/6 patients experience a DLT at any dose level except the highest dose level, 3 new patients will be enrolled at the next higher dose level; if 1/6 patients at the highest dose level experience a DLT, it will be deemed the MTD and the trial will stop. As soon as 2 patients experience a DLT at a given dose level, that dose will be concluded to be above the MTD, dose escalation will cease and 3 new patients will be enrolled at the next lower dose level. If 6 patients were previously treated at that lower dose, the study will halt and that lower dose will be declared the MTD. A subject who withdraws from the escalation phase of the study for reasons other than a DLT will be replaced.

FOLFIRINOX treatment will be given on Day 1 and 15 of the 4 weeks cycle and continued until unacceptable toxicity or disease progression, for a maximum of 12 cycles. Subjects will receive a single intravenous administration of Eryaspase on Day 1 and 15 of 4-weeks cycle.

The study visits are day 1, 8, 15, 22, during cycle 1 and day 1 and 15 during subsequent cycles with a 4-week follow-up period after the end of treatment. Subjects who show at least stable disease based on RECIST 1.1 at the end of the 12-week period (Day 85) are eligible for the continuation of FOLFIRINOX plus eryaspase treatment until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able to understand and willing to sign an IRB approved written informed consent document.
* Patient must have histologically or cytologically confirmed pancreatic adenocarcinoma, which is locally advanced, unresectable, or metastatic.
* Patient must have received no previous surgery, chemotherapy, radiotherapy or investigational therapy for the treatment of locally advanced or metastatic disease.
* If a patient has had adjuvant/neoadjuvant therapy for localized disease, tumor recurrence or disease progression must have occurred no sooner than 6 months after completing the last dose of the aforementioned therapies.
* Patient must have radiographically measurable disease according to RECIST 1.1
* Patient must be > 18 years of age.
* Patient must have a life expectancy of >= 3 months.
* Patient must have an ECOG performance status ≤ 1.
* Patient must have normal bone marrow and organ function as defined below:

  * Absolute neutrophil count >=1,500/mcl
  * Platelets >=100,000/mcl
  * Hemoglobin >=9.0 g/dL
  * Serum Albumin >=3.0 g/dL
  * Creatinine should be below the upper limit of normal OR Creatinine clearance (eGFR) >=60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
  * Plasma antithrombin III >= 65%, fibrinogen >= 150 mg/dL, international normalized ratio (INR) ≤ 1.5, and partial thromboplastin time (PTT) ≤ institutional ULN.
  * Total bilirubin ≤ 1.5x institutional ULN
* Patients who have had a stent placed for biliary obstruction can be included in the study.
* Female subject of childbearing potential must have a negative urine or serum pregnancy test.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Male subjects with a female partner of childbearing potential must agree to use two adequate methods or a barrier method plus a method of contraception

Exclusion Criteria:

* Evidence of neuroendocrine tumor, duodenal adenocarcinoma, or ampullary adenocarcinoma.
* History of other malignancy ≤ 3 years ago, with the exception of basal cell or squamous cell carcinoma of the skin, which were treated with local resection only or carcinoma in situ of the cervix of ductal carcinoma in situ.
* Receiving any other investigational agents 28 days prior to the screening process.
* Patient with evidence of brain metastases. Such patients must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to asparaginase, 5FU, oxaliplatin, or irinotecan.
* Any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection , symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, any clinically active malabsorption syndrome, inflammatory bowel disease, any condition that increases the risk of severe irinotecan gastrointestinal toxicity, or psychiatric illness/social situations that would limit compliance with study requirements
* Has an active autoimmune disease, or a documented history of autoimmune disease or syndrome that requires steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule.
* Has had an allogeneic tissue/solid organ transplant.
* Has received or will receive a live vaccine within 30 days prior to the first administration of study medication. Seasonal flu vaccines that do not contain live virus are permitted
* Has known active Hepatitis B or C.
* Patient is pregnant and/or breastfeeding.
* Known to be HIV-positive on combination antiretroviral.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus S Noel, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX: Eryaspase 75 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion).
  intravenous administration of mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
- Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX: Eryaspase 100 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion).
  intravenous administration of mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
- Eryaspase Dose Level -1 (50 Units/kg) Plus FOLFIRINOX: Eryaspase 50 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion).
  intravenous administration of mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
- Eryaspase Dose Level -2 (25 Units/kg) Plus FOLFIRINOX: Eryaspase 25 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion).
  intravenous administration of mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
Period: Overall Study
Arm/Group | Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX | Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX | Eryaspase Dose Level -1 (50 Units/kg) Plus FOLFIRINOX | Eryaspase Dose Level -2 (25 Units/kg) Plus FOLFIRINOX
Started | 3 | 16 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 16 | 0 | 0
Not completed — Physician Decision | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Progression of Disease | 2 | 5 | 0 | 0
Not completed — No Treatment per protocol | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX: Eryaspase (75 Units/kg) will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion)
  mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
- Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX: Eryaspase (100 Units/kg) will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion)
  mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
- Total: Total of all reporting groups
Arm/Group | Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX | Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX | Total
Number analyzed (Participants) | 3 | 16 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 8 | 9
  >=65 years | 2 | 8 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 1 | 8 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 2 | 15 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 2 | 8 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade 3 or 4 Adverse Events
Description: The number (percentage) of all subjects who experience Grad 3 or 4 treatment emergent adverse events (AEs), serious adverse events (SAEs), or abnormal laboratory results according to NCI CTCAE Version 5.0, that occur after Cycle 1, Day 1 will be reported until end of treatment visit.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX: Eryaspase 75 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion)
  mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
- Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX: Eryaspase 100 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion) in dose escalating/reduction depending on the cohort the patient is assigned to
  mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
Arm/Group | Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX | Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX
Number analyzed (Participants) | 3 | 16
Participants | 2 | 8

2. Secondary Outcome: Objective Response Rate by RECIST 1.1
Description: Number of participants with a complete or partial response from treatment as assessed by CT scan per RECIST 1.1 criteria.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX | Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX
Number analyzed (Participants) | 3 | 16
Participants | 1 | 3

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Time in months from start of treatment to disease progression, death, or completion of study which ever occurred first.
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX | Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX
Number analyzed (Participants) | 3 | 16
months | 5.6 [1.8 to 28.3] | 6.4 [0.4 to 34.7]

4. Secondary Outcome: Overall Survival (OS)
Description: The length of time from treatment initiation until death from any cause or off study date, whichever occurs first.
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX | Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX
Number analyzed (Participants) | 3 | 16
months | 10.2 [8.7 to 28.3] | 8.6 [0.4 to 34.7]

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed for 1 year (from Cycle 1, Day 1 will be reported until end of treatment visit.). All cause mortality was assessed up to 3 years.
Groups:
- Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX: Eryaspase 100 Units/kg will be administered on day 1 and 15 of a 4 week cycle (intravenous infusion)
  mFOLFIRINOX dosing will include 5-fluorouracil 2400 mg/m² over 46 hours, oxaliplatin 85 mg/m², Irinotecan 150 mg/m² (intravenous infusion) on Day 1 and 15 of the 4 weeks cycle for a maximum of 12 cycles.
Arm/Group | Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX | Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 3/3 | 13/16
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/16
Other Adverse Events (participants affected / at risk) | 3/3 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX (N=3) | Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX (N=16)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eryaspase Dose Level 0 (75 Units/kg) Plus FOLFIRINOX (N=3) | Eryaspase Dose Level 1 (100 Units/kg) Plus FOLFIRINOX (N=16)
Anemia (Blood and lymphatic system disorders) | 2 (6) | 11 (27)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Ear congestion
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (9)
Belching (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (10)
Diarrhea (Gastrointestinal disorders) | 2 (6) | 8 (21)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) — epigastric pain
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (2) | 8 (13)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (6)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (2) | 4 (6)
Fatigue (General disorders) | 2 (9) | 12 (35)
Fever (General disorders) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 2 (3) — Cold sensitivity
Generalized edema (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 8 (9)
Alkaline phosphatase increased (Investigations) | 3 (5) | 8 (10)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 6 (9)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 3 (5) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
GGT increased (Investigations) | 1 (1) | 5 (6)
Lipase increased (Investigations) | 1 (3) | 3 (3)
Neutrophil count decreased (Investigations) | 2 (5) | 3 (4)
Platelet count decreased (Investigations) | 2 (3) | 8 (13)
Serum amylase increased (Investigations) | 1 (3) | 2 (3)
Weight loss (Investigations) | 0 (0) | 3 (4)
White blood cell decreased (Investigations) | 2 (7) | 7 (9)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5) | 6 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (3)
Dysesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 4 (5)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 10 (19)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) — urinary abnormality-dysuria with frequency and urgency
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (3)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Hyperpigmentation of buccal mucosa
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (3)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT04292743/Prot_SAP_000.pdf